CLINICAL TRIAL: NCT03047967
Title: Effets du Tabagisme in Utero Sur la fonctionnalité de l'épithelium Respiratoire et Sur la Fonction Ventilatoire du Nouveau-né.
Brief Title: Effects of Prenatal Tobacco Smoke Exposure on Lung Function and Respiratory Epithelium Functionality in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C15-60
Record Dates: First submitted 2017-01-26; First posted 2017-02-09 (Estimated); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy Related; Tobacco Smoking; Lung Smokers; Newborn
MeSH Terms: conditions — Tobacco Smoking | interventions — Respiratory Function Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTSE (Experimental): Prenatal tobacco smoke exposed newborns. Lung function test Nasal brushing
  Interventions: Diagnostic Test: lung function tests; Diagnostic Test: Nasal brushing
- control (Experimental): Prenatal tobacco smoke non exposed newborns Lung function test Nasal brushing
  Interventions: Diagnostic Test: lung function tests; Diagnostic Test: Nasal brushing

INTERVENTIONS:
Diagnostic Test: lung function tests — baby-body plethysmography
Diagnostic Test: Nasal brushing — Epithelial sample collecting for in vitro study

SUMMARY:
Despite public campaigns to prevent cigarette smoking, it's about 20% of women who keep on smoking during pregnancy, exposing their fetus to prenatal tobacco adverse effects. Although environnemental tobacco smoke exposure effects are well known, consequences of prenatal tobacco smoke exposure (PTSE) need better caracterization. Previous animal study from our group have shown, in prenatal nicotine exposed mouse pups, alterations in tracheal epithelial structure similar to those observed in KO α7-nAChR mouse pups. These findings support the hypothesis that α7-nAChR are involved in the process of deleterious effects of tobacco smoking on respiratory epithelium development. The purpose of the present clinical study is to compare PTSE neonates with controls according to lung function and respiratory epithelial functionality. At the age of 3 days, small respiratory epithelium fragments will be obtained from gentle nasal brushing performed under antalgic premedication according to the method we previously published. Epithelium samples will be used for in vitro studies of α7-nAChR and CFTR functionality. Between the ages of 2 and 6 weeks, lung function testing will be performed, by means of baby-body plethysmography.

ELIGIBILITY:
Inclusion Criteria:

* inborn full-term neonate
* social security affiliation
* informed consent form signed by parents

Exclusion Criteria:

* prematurity < 35GW
* gemellary pregnancy
* Birth weight < 2200 g
* neonatal respiratory distress syndrome (nasal oxygenotherapy > 24 hours, invasive or noninvasive ventilation)
* neonatal malformation with conséquences on lung function
* neonatal liver or renal failure
* high risk of heritable lung disease
* contra-indication to saccharose or paracetamol antalgic use
* language barrier,
* mother refusal to declare or precise her tobacco consumption
* no social security cover
* informed consent form not signed

Ages: 2 Days to 6 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2019-02-09 (Actual)

PRIMARY OUTCOMES:
α7-nAChR functionnality | day 3
  calcium influx mesurements on epithelial fragments by monitoring changes in Fluo-4 fluorescence intensity.
  Fluo-4 is a fluorescent dye which fluorescence is modified by its linkage to Calcium. Its fluorescence changes measurements shows calcium cellular flows.
CFTR functionality | day 3
  chlorid influx study on epithelial fragmentsby monitoring changes in spq fluorescence intensity.
  sqp is a fluorescent dye which fluorescence is modified by its linkage to Chlore. Its fluorescence changes measurements shows chlore cellular flows.

SECONDARY OUTCOMES:
Lung function test | between ages 2 and 6 week
  baby-body plethysmography that study ventilation in asleep infants (measurement of tidal volumes, respiratory frequency, airway resistances, respiratory system compliance, maximal expiratory flows)
ciliary frequency mesurement | day 3
  On epithelial fragments. By using vidéo microscopy and select several delimited zone where ciliary frequency is measured. Then a mean freqeuncy is calculated

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MAURAN, MD PHD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Inserm, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided